CLINICAL TRIAL: NCT05146128
Title: Functional or Analytic Methods: What is the Best to Strengthen Shoulder and Scapular Muscles?
Brief Title: Comparison Between Functional and Analytic Methods to Strengthen Shoulder Rotators and Scapular Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Camille Tooth, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Functional or analytic
Record Dates: First submitted 2021-11-09; First posted 2021-12-06 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Strength

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were allocated to a group in a random way
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Analytic group (Experimental): The participants had to perform analytic exercices for shoulder rotators and scapular stabilizing muscles
  Interventions: Other: Strengthening exercises
- Functional group (Experimental): The participants had to perform functional exercices for shoulder rotators and scapular stabilizing muscles
  Interventions: Other: Strengthening exercises
- Mixed group (Experimental): The participants had to perform both analytic and functional exercices for shoulder rotators and scapular stabilizing muscles
  Interventions: Other: Strengthening exercises

INTERVENTIONS:
Other: Strengthening exercises — The participants had to perform specific exercices 3 times a week during 8 weeks

SUMMARY:
The objective of the study was to compare analytic, functional and mixed (analytic/functional) methods in strengthening rotator cuff and scapular stabilizers muscles. For that purpose, participants had to follow a strengthening program 3 times a week during 8 weeks.

DETAILED DESCRIPTION:
Each participant was allocated to a group (analytic, functional and mixed groups) in a random way while assuring that the groups were quite similar in morphological data or in performance. The strengthening program has to be performed three times a week during eight weeks by each participant.

The exercises included in the program were chosen among the bests exercises described in literature to active shoulder rotators as well as scapular stabilizing muscles. The analytic group has to perform the following exercises: prone rowing with dumbbell, prone external rotation at 90° of abduction, prone extension, bilateral scapular protraction with dumbbells, eccentric internal rotation at 90° of abduction, external rotation diagonal exercise and single arm shot put medicine ball throw. The functional group performed the same exercises but with a functional component: standard plank rowing, swissball external rotation at 90° of abduction, standard plank extension, bilateral scapular protraction (standard plank + raised feet), eccentric internal rotation 90° of abduction with unipodal glute bridge, external rotation diagonal in an unipodal position and single arm shot put throw with medicine ball in and single arm shot put medicine ball throw. Then, for the mixed group, the program included exercises from the analytic group and other ones from the functional group in equal parts. For all the groups, the exercises aimed to strengthen shoulder rotators were performed five times in a row and the others aimed to strengthen scapular stabilizing muscles were performed fifteen times in a row. The only exception was for the single arm shot put medicine ball throw that was performed ten times. Two series of each exercises were performed during each session, which represent a mean duration of thirty minutes.

At the beginning and at the end of the intervention, three different evaluations were performed :

* Measurement of shoulder rotators strength (with an isokinetic device)
* Measurement of scapular stabilizers strength (with an isokinetic device)
* Measurement of functional performance (with Medicine Ball Throw, CKCUEST, Y Balance Test and a core stability test)

ELIGIBILITY:
Inclusion Criteria:

* Males aged between 18 and 35 years old

Exclusion Criteria:

* Practicing an overhead sport
* Having an history of shoulder pain or shoulder surgery in the past 12 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Shoulder rotators strength | Change from baseline at 8 weeks
  The strength was measured with an isokinetic device
Scapular stabilizing muscles strength | Change from baseline at 8 weeks
  The strength was measured with an isokinetic device
Upper Quarter Y Balance Test | Change from baseline at 8 weeks
  A closed-kinetic-chain upper extremity functional test aimed to assess stability and mobility of the shoulder
Closed Kinetic Chain Upper Extremity Stability Test | Change from baseline at 8 weeks
  A closed-kinetic-chain upper extremity functional test aimed to assess coordination and shoulder stability
Medicine ball throw | Change from baseline at 8 weeks
  The participants had to throw a 800g-medicine ball as far as possible
Core stability test | Change from baseline at 8 weeks
  The participants had to maintain a plank position as long as possible

CONTACTS AND LOCATIONS:
Overall Officials: Camille Tooth, Principal Investigator — ULiège
Locations (1):
- Université de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No